CLINICAL TRIAL: NCT06201676
Title: Low-Dose Short-Term Ketorolac to Reduce Chronic Opioid Use in Orthopaedic Polytrauma Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Arun Aneja, MD, PhD, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023P003287; HT9425-23-1-0413 (Other Grant/Funding Number: Department of Defense PRORP)
Record Dates: First submitted 2023-12-16; First posted 2024-01-11 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Orthopaedic Polytrauma; Chronic Opioid Use
Keywords: orthopaedic polytrauma; chronic opioid use; NSAID; IV ketorolac; acute pain management
MeSH Terms: interventions — Ketorolac; Ketorolac Tromethamine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Parallel, two-arm, placebo-controlled, randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participants, their primary treatment teams, study investigators, research personnel, and the statistician will be blinded to each participant's group assignment. A central randomization scheme will be created by the statistician and provided to the Clinical Trials Pharmacy at both sites. Clinical Trials Pharmacy will be the only stakeholders in this study who will be unmasked to the participant's group assignment. The statistician will be blinded to each subject's group assignment when provided with the final dataset for analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard of Care (SOC) + Ketorolac (Experimental): The treatment arm will receive 15 mg of intravenous (IV) ketorolac every 6 hours during the first five hospital days, in addition to standard of care (SOC) multimodal analgesia according to each site's institutional protocol.
  Interventions: Drug: Ketorolac Injection
- Standard of Care (SOC) (Placebo Comparator): The placebo arm will receive 2 mL of intravenous (IV) saline every 6 hours during the first five hospital days, in addition to standard of care (SOC) multimodal analgesia according to each site's institutional protocol.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: Ketorolac Injection — Ketorolac tromethamine is a nonsteroidal anti-inflammatory drug (NSAID) that exhibits analgesic activity in animal models. The mechanism of action of ketorolac, like that of other NSAIDs, is not completely understood but may be related to prostaglandin Reference ID: 3281582 3 synthetase inhibition. The biological activity of ketorolac tromethamine is associated with the S-form. Ketorolac tromethamine possesses no sedative or anxiolytic properties.
  Other Names: Toradol
  Arms: Standard of Care (SOC) + Ketorolac
Other: Normal Saline — 0.9% Sodium Chloride Injection, USP is sterile and nonpyrogenic. It is a parenteral solution containing sodium chloride in water for injection intended for intravenous administration. Each 100 mL of 0.9% Sodium Chloride Injection, USP contains 900 mg sodium chloride in water for injection. Electrolytes per 1000 mL: sodium (Na+) 154 mEq; chloride (Cl-) 154 mEq. The osmolarity is 308 mOsmol/L (calc.).
  Other Names: Sodium Chloride
  Arms: Standard of Care (SOC)

SUMMARY:
The goal of this randomized clinical trial is to learn if the use of a low-dose nonsteroidal anti-inflammatory drug (NSAID), ketorolac, reduces the rate of chronic opioid use in orthopaedic polytrauma patients. The main questions this study aims to answer are:

1. Are patients who are given scheduled ketorolac during the first five hospital days less likely to develop chronic opioid use at 6 months after injury compared to patients who receive placebo?
2. Does scheduled ketorolac during the first five hospital days improve functional responses to pain at discharge, 3 months, and 6 months after injury?
3. Does early pain control provided by ketorolac decrease chronic opioid use through decreased acute pain and opioid use, improved functional responses to pain, or both?

Participants will be enrolled and randomized to either the ketorolac (treatment) group or placebo group to be given every 6 hours during the first five hospital days. Pain and opioid use will be measured daily during the five-day treatment period. Opioid use will be measured and functional response to pain surveys will be obtained at discharge, 2 weeks, 6 weeks, 3 months, and 6 months after injury.

Researchers will compare ketorolac (treatment) versus saline (placebo) to see if ketorolac reduces chronic opioid use and improves the functional response to pain.

DETAILED DESCRIPTION:
Background: Post-traumatic pain (PTP) can be difficult to control in polytrauma patients. Currently, opioids serve as the cornerstone for pain management despite their potential for complications including chronic use. Given this, it is not surprising that new-onset opioid abuse is a leading cause of complications following polytrauma and can be a limiting factor in delaying and/or safely resuming pre-injury responsibilities. Changes in pain management are needed to help military personnel and civilians expeditiously and safely return to their pre-injury duty. Early short-term scheduled ketorolac treatment has been shown to decrease acute pain and short and mid-term opioid use but whether this translates into decreased chronic opioid use is unknown.

Hypothesis/Objective: This study attempts to determine whether an early scheduled short-term course of ketorolac treatment has a sustained impact by decreasing chronic opioid use. The study will also investigate whether this treatment improves function and resilience as well as whether early pain control and/or the functional response to pain mediate (i.e. are responsible for / explain) the effect of the ketorolac intervention on chronic opioid use.

Specific Aims:

Aim 1: Determine whether orthopaedic polytrauma patients who receive IV ketorolac, 15 mg every six hours, in combination with standard of care (SOC) analgesia for the first five inpatient days are less likely to develop chronic opioid use, defined as continued use at six months post-injury, compared to patients receiving similar placebo injections in combination with SOC.

Aim 2: Determine if patients who received a consistent five-day course of low-dose ketorolac during the inpatient stay have an improved functional response to pain measured via: 1) Brief Pain Inventory (BPI), 2) Patient-Reported Outcomes Measurement Information System - Pain Interference (PROMIS-PI), and 3) Brief Resilience Scale (BRS) scores at discharge, 3 months, and 6 months post-injury. Secondary pain outcome measures such as pain VAS and MME data will also be compared between the two groups.

Aim 3: Determine (1) the extent to which early pain control during the intervention, assessed using pain VAS and MME intake, mediates the effect of ketorolac on chronic opioid use, (2) the extent to which early pain control mediates the effect of ketorolac on the functional response to pain measures, assessed using BPI, PROMIS-PI, and BRS, and (3) the extent to which early pain control and the functional response to pain in combination or isolation mediate the effect of ketorolac on chronic opioid use.

Study Design: Polytrauma patients aged 18 to 70 years of age with a New Injury Severity Score greater than 9, consistent with moderate injury, and anticipated admission of at least 5 days to ensure completion of the treatment will be enrolled. Once enrolled, patient randomization will be stratified by site and NISS score categorization (either 10-15 or greater than 15). Experienced clinical research staff will prospectively identify patients with strict adherence to all inclusion and exclusion criteria. Participants will be randomized to treatment (15 mg of ketorolac plus SOC multimodal analgesia every 6 hours for 5 days) or control (similar volume of saline every 6 hours plus SOC multimodal analgesia for 5 days). Measures of the functional response to pain including the BPI, PROMIS-PI, and BRS will be collected at hospital discharge and 3- and 6-months post-injury. Outcome measures of pain including VAS and MME will be recorded at enrollment, during the first five days of inpatient admission, at discharge, and at clinic follow-ups. The treatment and control groups will be compared using the intention-to-treat analyses across the primary and secondary outcomes. Mediation analyses will be used to understand how early pain control and the functional response to pain mediate the effect or lack of effect on chronic opioid use to better understand the factors that lead to this devastating complication.

ELIGIBILITY:
Inclusion Criteria:

* Patient age: 18-70
* Patient or legally authorized representative (LAR) able to provide consent
* Patients with NISS ≥ 9 at time of admission with musculoskeletal trauma requiring surgical fixation
* Anticipated admission ≥ 5 days
* Patients who speak English or Spanish
* Patients who can be followed at the enrolling facility for at least 6 months

Exclusion Criteria:

* Patient age < 18 or > 70 years
* Patients with injury more than 24 hours prior to evaluation
* Patients with active hemorrhagic shock or risk of significant hemorrhage
* Patients who are pregnant or breastfeeding
* Patients with a history of active gastrointestinal bleeds or ulceration
* Patients with chronic use of steroids or immune-modulating drugs or history of organ transplantation
* Patients with preexisting chronic renal, liver, heart, or lung disease
* Patients with a creatinine ≥ 1.30 mg/dL during enrollment
* Patients with history of myocardial infarction, stroke, or bleeding disorder
* Patients with head or chest injury requiring surgical intervention
* Patients with allergy to ketorolac or hypersensitivity to aspirin
* Patients receiving chronic opioid therapy or treatment for opioid use disorder
* Patients who are current IV drug users
* Patients who require a daily NSAID or aspirin regimen, except for daily low-dose aspirin (81 mg)
* Patients with insufficient follow-up or anticipated difficulty in completing follow-up at a study site for a minimum of 6 months due to any of the follow reasons: death, no follow-up after initial discharge, severe psychiatric conditions, unstable living conditions, planned follow-up at another medical center not participating in this study, live far away from the clinic, and/or incarcerated

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Chronic Opioid Use | 6 months
  Defined as continued opioid use at 6 months post-trauma

SECONDARY OUTCOMES:
Brief Pain Inventory (BPI) | Enrollment, Hospital Discharge (up to 2 weeks), 2 weeks, 6 weeks, 3 months, and 6 months post-trauma
  Pain assessment tool that measures both the intensity of pain and interference of pain in a patient's life, including pain relief, pain quality, and patient perception of pain. Each question is scaled from 0 to 10, with a higher score meaning worse pain.
Patient-Reported Outcomes Measurement Information System-Pain Interference (PROMIS-PI) | Hospital Discharge (up to 2 weeks), 2 weeks, 6 weeks, 3 months, and 6 months post-trauma
  NIH-validated outcome measure that assesses how pain interferes with a patient's daily activities. This is measured using a T-score metric in which 50 is the mean of a relevant reference population, and 10 is the standard deviation of the population. A higher score for this survey means a worse outcome and is representative of pain interfering more in a patient's daily activities.
Brief Resilience Scale (BRS) | Hospital Discharge (up to 2 weeks), 2 weeks, 6 weeks, 3 months, and 6 months post-trauma
  Scale developed to assess a patient's ability to bounce back or recover from stress. This scale consists of 6 questions with answer choices ranging from 1-5. The total score is calculated and averaged to reflect the BRS score. BRS scores from 1.00 - 2.99 reflect low resilience, 3.00 - 4.30 reflect normal resilience, and scores from 4.31 - 5.00 reflect high resilience.
Visual Analogue Scale (VAS) | Enrollment, First Five Hospital Days, Hospital Discharge (up to 2 weeks), 2 weeks, 6 weeks, 3 months, and 6 months post-trauma
  Instrument that attempts to capture a patient's perception of pain along a continuum. This will be measured on a scale of 0 - 100, with 0 being no pain, 50 being moderate pain, and 100 being the worst pain possible.
Morphine Milligram Equivalents (MME) | Enrollment, First Five Hospital Days, Hospital Discharge (up to 2 weeks)
  Calculation used to standardize opioid consumption.
Opioid Use | 2 weeks, 6 weeks, 3 months, and 6 months post-trauma
  A survey to assess if patients are using opioids in the outpatient setting

CONTACTS AND LOCATIONS:
Overall Officials: Arun Aneja, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Pilot Study Results — https://journals.lww.com/jorthotrauma/fulltext/2023/12000/low_dose_short_term_scheduled_ketorolac_reduces.7.aspx
- See also: Pilot Study Results #2 — https://journals.lww.com/jorthotrauma/abstract/9900/does_scheduled_low_dose_short_term_nsaid.357.aspx